CLINICAL TRIAL: NCT06965959
Title: THE EFFECT OF EXERGAMING APPLICATION AND AUTOGENIC RELAXATION TECHNIQUE ON PSYCHOLOGICAL WELL-BEING AND LIFE ENGAGEMENT OF NURSING HOME RESIDENTS
Brief Title: THE EFFECT OF EXERGAMING APPLICATION AND AUTOGENIC RELAXATION TECHNIQUE ON PSYCHOLOGICAL WELL-BEING AND LIFE ENGAGEMENT OF NURSING HOME RESIDENTS: A RANDOMİZED CONTROLLED TRİAL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cumhuriyet University (Other)
Responsible Party: Principal Investigator, Mehtap Budak, PhD Student in Nursing, Cumhuriyet University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2023-04/50
Record Dates: First submitted 2025-05-02; First posted 2025-05-11 (Actual); Last update posted 2025-05-11 (Actual); Status verified 2025-05

CONDITIONS: Psychological Well-being; Nursing Homes Residents; Aging; Exergaming; Mind-Body Therapies; Quality of Life; Health Promotion
Keywords: Exergaming; Autogenic Relaxation; Psychological Well-Being; Life Engagement; Nursing Home Residents
MeSH Terms: conditions — Psychological Well-Being | interventions — Autogenic Training

STUDY DESIGN:
Intervention Model Description: Participants were randomly assigned to one of three parallel groups: (1) exergaming intervention group, (2) autogenic relaxation intervention group, and (3) control group. Each group received their assigned intervention separately, and no crossover occurred between arms.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Exergaming Intervention Group (Experimental): Participants in this group engaged in exergaming sessions using motion-based digital games (e.g., table tennis, boxing, skiing) twice per week for 8 weeks.
  Interventions: Behavioral: Exergaming Intervention Group
- Autogenic Relaxation Intervention Group (Experimental): Participants in this group practiced autogenic relaxation twice per week for 8 weeks in small groups guided by verbal instructions
  Interventions: Behavioral: Autogenic Relaxation
- Control Group (No Intervention): Participants in this group received no intervention and continued their usual routine.

INTERVENTIONS:
Behavioral: Exergaming Intervention Group — A behavioral intervention involving the use of motion-based digital games such as table tennis, boxing, skiing, and bowling. Participants performed exergaming sessions twice per week for eight weeks. Each session lasted approximately 15 minutes and was conducted in pairs under supervision. The intervention aimed to promote physical activity, cognitive engagement, and social interaction among older adults in a nursing home setting.
  Arms: Exergaming Intervention Group
Behavioral: Autogenic Relaxation — A behavioral mind-body intervention in which participants practiced standardized verbal relaxation techniques focused on passive concentration and bodily awareness. Sessions were conducted in quiet rooms in small groups, twice per week for eight weeks, each lasting approximately 15 minutes. The goal was to enhance psychological well-being and reduce emotional tension in institutionalized older adults.
  Arms: Autogenic Relaxation Intervention Group

SUMMARY:
This interventional clinical trial was conducted to evaluate the effects of Antroyun (exergaming) and autogenic relaxation techniques on psychological well-being and life engagement among older adults living in nursing homes. Participants were randomly assigned to one of three groups: Antroyun intervention group, autogenic relaxation group, and a control group. Interventions were applied twice per week for eight weeks.

The results indicated that both interventions had a significant effect on improving psychological well-being and life engagement. The Antroyun group showed faster and more marked improvements in earlier follow-ups, while the autogenic relaxation group demonstrated sustained benefits in later follow-ups. The control group did not show any significant changes over time. Additionally, in the Antroyun group, the number of game wins was positively correlated with improvements in psychological well-being and life engagement scores.

This study was carried out as part of a doctoral dissertation at Sivas Cumhuriyet University.

DETAILED DESCRIPTION:
This study was registered retrospectively due to its nature as a doctoral dissertation and institutional administrative timelines. Although participant enrollment and data collection had already started, the study protocol and outcome measures were pre-specified and ethically approved prior to implementation. No interim analysis was conducted prior to registration. This registration is intended to enhance research transparency and integrity.

ELIGIBILITY:
Inclusion Criteria:

* Age 65 years or older
* Residing in a nursing home
* Able to communicate and follow instructions
* Scoring 24 or above on the Standardized Mini Mental Test (SMMT)
* Voluntary participation and written informed consent obtained

Exclusion Criteria:

* Diagnosed with advanced cognitive impairment (SMMT score < 24)
* Diagnosed with severe psychiatric disorders (e.g., schizophrenia, severe depression)
* Having physical disabilities that prevent participation in the interventions (e.g., immobility, severe visual or auditory loss)
* Refusal or inability to provide informed consent

Ages: 65 Years to 95 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 69 (Actual)
Dates: Start 2024-02-01 (Actual); Primary Completion 2024-08-01 (Actual); Study Completion 2024-08-01 (Actual)

PRIMARY OUTCOMES:
Change in Psychological Well-Being Score | Baseline, Week 4, Week 8, and Week 16 (4 follow-ups total)
  Psychological well-being was measured using the Elderly Psychological Well-Being Scale. The scale evaluates emotional, cognitive, and social well-being. Higher scores indicate better psychological well-being.
Change in Life Engagement Score | Baseline, Week 4, Week 8, and Week 16 (4 follow-ups total)
  Life engagement was assessed with the Life Engagement Scale for Older Adults, which measures the degree of purpose, activity, and connectedness perceived by the elderly.
Standardize Mini Mental Test | Baseline
  Cognitive function was evaluated using the Standardized Mini Mental Test (SMMT), which assesses orientation, registration, attention, recall, and language. The test was used to monitor cognitive stability during the study.

CONTACTS AND LOCATIONS:
Locations (1):
- Sivas Cumhuriyet University, Institute of Health Sciences, Sivas, Central, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided